CLINICAL TRIAL: NCT02621203
Title: Investigate to Medications, Re-hospitalization and Mortality of Patients With Hospitalized Acute Heart Failure Patients
Brief Title: Patient Journey in Hospital With Acute Heart Failure
Acronym: JourneyHF-TR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mehdi Zoghi (Other)
Responsible Party: Sponsor-Investigator, Mehdi Zoghi, Prof., Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital
Organization: Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital (Other)
Other Study IDs: Cardiovascular Academy
Record Dates: First submitted 2015-11-16; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A multicentre, prospective, observational, hospital-based registry of patients with acute heart failure (AHF) those whose care was guided by a cardiologist in Turkey.

DETAILED DESCRIPTION:
The purpose of this study is to compose a national database of the etiologies, clinical and demographic characteristics, using diagnostic tests, precipitating and risk factors, management of from intensive care unit (ICU) or coronary care unit to hospital discharge, length of stay in the ICU and hospital, in-hospital mortality and discharge medications of hospitalized AHF patients in Turkish population.

The etiologies, precipitating factors, demographics, clinical characteristics, management and outcome of patients admitted in hospital with acute heart failure in Turkish population will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* Clinical diagnosis of acute heart failure
* Admitted to the participating hospitals

Exclusion Criteria:

* Patients <18 years old
* Patients with acute heart failure who are discharged from the emergency room without admission.
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital-based registry of patients with acute heart failure (AHF) those whose care was guided by a cardiologist in Turkey.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 3 months

SECONDARY OUTCOMES:
Hospitalization | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Zoghi, MD, Study Director — mehdi_zoghi@hotmail.com
Locations (1):
- Dr. Ahmet ekmekçi, Istanbul, Turkey (Türkiye)